

# **Trial Statistical Analysis Plan**

c21117747-01

| BI Trial No.: | 1305-0020 |
|---|---|
| Title: | Relative bioavailability of BI 1015550 following oral administration under fed and fasted conditions in healthy male subjects |
| Investigational Products: | BI 1015550 |
| Responsible trial statisticians: | |
| | Phone:<br>Fax: |
| | Phone:<br>Fax: |
| Date of statistical analysis plan: | 19 JAN 2018 SIGNED |
| Version: | "Final" |
| Proprietary confidential information © 2018 Boehringer Ingelheim International GmbH or one or more of its affiliated companies. All rights reserved | |

This document may not - in full or in part - be passed on, reproduced, published or otherwise used without prior written permission.

TSAP for BI Trial No: 1305-0020 

Proprietary confidential information © 2018 Boehringer Ingelheim International GmbH or one or more of its affiliated companies

#### 1. TABLE OF CONTENTS

| TITLE | PAGE | 1 |
|----------------|------------------------------------------------|-----------|
| 1. | TABLE OF CONTENTS | 2 |
| LIST O | OF TABLES | 4 |
| 2. | LIST OF ABBREVIATIONS | 5 |
| 3. | INTRODUCTION | 7 |
| 4. | CHANGES IN THE PLANNED ANALYSIS OF THE STUDY | |
| 5. | ENDPOINTS PRIMARY ENDPOINTS | |
| 5.1 | | |
| 5.2 | SECONDARY ENDPOINTS | |
| 5.2.1 | Key secondary endpoints | |
| 5.2.2 | Secondary endpoints | |
| <b>6.</b> | GENERAL ANALYSIS DEFINITIONS | 11 |
| 6.1 | TREATMENTS | |
| <b>6.2</b> | IMPORTANT PROTOCOL VIOLATION | 12 |
| 6.3 | PATIENT SETS ANALYSED | 14 |
| | | 15 |
| 6.5 | POOLING OF CENTRES | |
| 6.6 | HANDLING OF MISSING DATA AND OUTLIERS | |
| <b>6.7</b> | BASELINE, TIME WINDOWS AND CALCULATED VISITS | |
| 7. | PLANNED ANALYSIS | |
| <b>7.1</b> | DEMOGRAPHIC AND OTHER BASELINE CHARACTERISTICS | |
| <b>7.2</b> | CONCOMITANT DISEASES AND MEDICATION | 18 |
| 7.3 | TREATMENT COMPLIANCE | |
| <b>7.4</b> | PRIMARY ENDPOINTS | |
| 7.5 | SECONDARY ENDPOINTS | <b>20</b> |
| 7.5.1 | Key secondary endpoints | <b>20</b> |
| 7.5.2 | Secondary endpoints | |
| 7.7 | EXTENT OF EXPOSURE | |
| 7.7<br>7.8 | SAFETY ANALYSIS | |
| 7.8.1 | Adverse events. | |
| 7.8.2 | Laboratory data | |
| 7.8.2<br>7.8.3 | Vital signs | |
| 7.8.4 | ECG. | |
| 7.8.5 | Others | |
| 8. | REFERENCES | |
| | , | <b>26</b> |

| Boehringer Ingelheim |
|---------------------------------|
| TSAP for BI Trial No: 1305-0020 |

| <b>Page</b> | 3 | of | 27 |
|-------------|---|----|----|

| Proprietary co | onfidential information © 2018 Boehringer Ingelheim International GmbH | or one or more of its affiliated companies |
|---|---|---|
| 10. | HISTORY TABLE | 27 |

## **Boehringer Ingelheim**

TSAP for BI Trial No: 1305-0020 

Proprietary confidential information © 2018 Boehringer Ingelheim International GmbH or one or more of its affiliated companies

## LIST OF TABLES

| Table 6.1: 1 | Treatments and labels used in the analysis | 11 |
|--------------|--------------------------------------------|----|
| | Important protocol violations | |
| | Subject sets analysed | |
| | History table | |
| | === <i>J</i> | |

TSAP for BI Trial No: 1305-0020 

Proprietary confidential information © 2018 Boehringer Ingelheim International GmbH or one or more of its affiliated companies

#### 2. LIST OF ABBREVIATIONS

| Term | Definition / description |
|---|---|
| ADS | Analysis dataset |
| AE | Adverse event |
| AESI | Adverse event of special interest |
| ALT | Alanine aminotransferase |
| ANOVA | Analysis of variance |
| AST | Aspartate aminotransferase |
| $AUC_{0\text{-tz}}$ | Area under the concentration-time curve of the analyte in plasma over the time interval from 0 to the last quantifiable data point |
| $AUC_{0-\infty}$ | Area under the concentration-time curve of the analyte in plasma over the time interval from 0 extrapolated to infinity |
| BI | Boehringer Ingelheim |
| BMI | Body mass index |
| BWC | Bioavailability/Bioequivalence, within-subject design, time-controlled |
| $C_{max}$ | Maximum measured concentration of the analyte in plasma |
| CTP | Clinical Trial Protocol |
| CTR | Clinical Trial Report |
| CV | Arithmetic coefficient of variation |
| DBLM | Database lock meeting |
| DILI | Drug induced liver injury |
| ECG | Electrocardiogram |
| EudraCT | European Union Drug Regulating Authorities Clinical Trials |
| gCV | Geometric coefficient of variation |
| gMean | Geometric mean |
| ICH | International Conference on Harmonisation |
| ISF | Investigator site file |
| LLT | Lower level term |
| Max | Maximum |
| MedDRA | Medical Dictionary for Regulatory Activities |
| Min | Minimum |
| N | Number non-missing observations |

TSAP for BI Trial No: 1305-0020 

Proprietary confidential information © 2018 Boehringer Ingelheim International GmbH or one or more of its affiliated companies

| Term | Definition / description |
|---|---|
| O*C | Oracle Clinical |
| PD | Pharmacodynamic(s) |
| PK | Pharmacokinetic(s) |
| PKS | PK parameter set |
| PT | Preferred term |
| PV | Protocol violation |
| qd | Quaque die (daily) |
| R | Reference treatment |
| RAGe | Report Appendix Generator system |
| REP | Residual effect period |
| RPM | Report planning meeting |
| $\mathrm{SAS}^{\circledR}$ | Statistical Analysis System |
| SD | Standard deviation |
| SOC | System organ class |
| T | Test treatment |
| $t_{max}$ | Time from dosing to maximum measured concentration of the analyte in plasma |
| TS | Treated set |
| TSAP | Trial statistical analysis plan |
| ULN | Upper limit of normal |
| WHO-DD | World Health Organization Drug Dictionary |
| XPKISTAT | Library of SAS® Macros for PK analysis |

TSAP for BI Trial No: 1305-0020

Proprietary confidential information © 2018 Boehringer Ingelheim International GmbH or one or more of its affiliated companies

### 3. INTRODUCTION

As per ICH E9 (1), the purpose of this document is to provide a more technical and detailed elaboration of the principal features of the analysis described in the protocol, and to include detailed procedures for executing the statistical analysis of the primary and secondary variables and other data.

This Trial statistical analysis plan (TSAP) assumes familiarity with the Clinical Trial Protocol (CTP). In particular, the TSAP is based on the planned analysis specification as written in CTP Section 7 "Statistical Methods and Determination of Sample Size". Therefore, TSAP readers may consult the CTP for more background information on the study, e.g., on study objectives, study design and population, treatments, definition of measurements and variables, planning of sample size, randomisation.

Study data will be stored in a trial database within the Oracle ClinicalTM (O\*C) system.

Pharmacokinetic (PK) parameters will be calculated using Phoenix WinNonlin<sup>TM</sup> software (version 6.3, Certara USA Inc., Princeton, NJ, USA).

The statistical analyses will be performed within the validated working environment CARE, including SAS<sup>®</sup> (current Version 9.4, by SAS Institute Inc., Cary, NC, USA), and a number of SAS<sup>®</sup>-based tools (e.g., macros for the analyses of AE data or laboratory data; Report Appendix Generator system (RAGe) for compilation/formatting of the CTR appendices).

### 4. CHANGES IN THE PLANNED ANALYSIS OF THE STUDY

All analyses as planned in the CTP will be performed and are described in more detail in this TSAP. The following change compared to the protocol will be made:

No 'Entered set' will be defined in the TSAP as data of subjects entered and randomised but discontinued before first administration of trial medication will not be entered in the case report form. A correct display of the 'Entered set' would not be possible.

TSAP for BI Trial No: 1305-0020

Proprietary confidential information © 2018 Boehringer Ingelheim International GmbH or one or more of its affiliated companies

### 5. ENDPOINTS

### 5.1 PRIMARY ENDPOINTS

**Section 5.5.1.1 of the CTP:** *The following primary endpoints will be determined for BI 1015550:* 

- $AUC_{0-tz}$  (area under the concentration-time curve of the analyte in plasma over the time interval from 0 to the last quantifiable data point)
- $C_{max}$  (maximum measured concentration of the analyte in plasma)

#### 5.2 SECONDARY ENDPOINTS

### 5.2.1 Key secondary endpoints

This section is not applicable as no key secondary endpoints have been defined in the CTP.

### 5.2.2 Secondary endpoints

**Section 5.5.1.2 of the CTP:** *The following secondary endpoint will be evaluated for BI 1015550:* 

•  $AUC_{0-\infty}$  (area under the concentration-time curve of the analyte in plasma over the time interval from 0 extrapolated to infinity)

TSAP for BI Trial No: 1305-0020 

Proprietary confidential information © 2018 Boehringer Ingelheim International GmbH or one or more of its affiliated companies

### 6. GENERAL ANALYSIS DEFINITIONS

#### 6.1 TREATMENTS

For basic study information on investigational products, assignment of treatment sequences and selection of doses, please see CTP, Sections 3 and 4.

The study will be performed as a randomised, open-label, single dose, two-way crossover trial with 2 treatments (T and R) and 2 treatment sequences (TR or RT).

In total, it was planned to assign 12 healthy male subjects to the two treatment sequences in a 1:1 ratio.

For details of dosage and formulation see <u>Table 6.1: 1</u> below:

Table 6.1: 1 Treatments and labels used in the analysis

| Treatment | | Short label |
|-----------|---------------------------------------|--------------|
| T | BI 1015550, 4*6 mg tablet, fed, qd | BI 24mg fed |
| R | BI 1015550, 4*6 mg tablet, fasted, qd | BI 24mg fast |

The following separate study phases will be defined for the analyses of AEs:

- Screening (ranging from 0:00 h on day of informed consent until first administration time of study drug)
- On treatment (including residual effect period (REP); i.e. ranging from the time of administration of the respective treatment until thereafter)
- Follow-up (ranging from end of on treatment phase until next drug administration or 0:00 h on the day after trial termination date, according to previous treatment (labelled "FU-Test", "FU-Ref"))

Displays of AEs will be presented separately for the treatments described in Table 6.1: 1 above.

Two types of AE displays will be provided in the report:

A) Section 15.3 and Appendix 16.1.9.2.8 (for ClinicalTrials.gov and EudraCT only) of the CTR displays:

In these displays, the on treatment phase will be analysed (labelled with the name of the study treatment (short label)). Screening and follow-up periods will not be included in this analysis. The following total will be provided in addition (Section 15.3 only):

• a total over all on treatment phases included in this analysis ("Total on treatment")

B) Section 15.4 and Appendix 16.1.9.2.8 (except for ClinicalTrials.gov and EudraCT) of the CTR displays:

- Screening
- On treatment (labelled with the name of the study treatment (short label))
- Follow-up ("FU-Test" and "FU-Ref")

In Section 16.1.9.2.8 AE tables, the following totals will be provided in addition:

• a total over all study phases ("**Total**")

Tables of vital signs and laboratory values will present results by the above mentioned on treatment phase.

For detailed information on the handling of the treatments in the O\*C views refer to Technical TSAP ADS plan. In particular, AEs will be counted for test or reference treatment if they occur up to the end of the residual effect period

#### 6.2 IMPORTANT PROTOCOL VIOLATION

Data discrepancies and deviations from the CTP will be identified for all randomised subjects. Listings of protocol deviations and of unresolved discrepancies will be provided to be discussed at the combined report planning and database lock meeting (RPM/DBLM), e.g. deviations in drug administration, in blood sampling etc. At this meeting, it will be decided whether the discrepant data can be used as they are or whether the data have to be corrected in the clinical database.

Each protocol deviation must be assessed to determine whether it is an important protocol violation. A protocol violation (PV) is important if it affects the rights or safety of the study subjects or if it can potentially influence the primary outcome measure(s) for the respective subjects in a way that is neither negligible nor in accordance with the study objectives. This last category of important PV forms the basis for the decision of whether a subject does or does not belong to an analysis set. PVs that do not influence the subject's rights and safety or the evaluability of the subjects for the main study objectives are called non-important PVs. These are only considered when checking the trial quality in general.

If any important PVs are identified, they are to be summarised into categories and will be captured in the RPM/DBLM minutes via an accompanying Excel spreadsheet [001-MCS-50-413\_RD-02] (2). The following table contains the categories which are considered to be important protocol violations in this trial. If the data show other important PVs, this table will be supplemented accordingly by the time of the RPM/DBLM.

TSAP for BI Trial No: 1305-0020 

Proprietary confidential information © 2018 Boehringer Ingelheim International GmbH or one or more of its affiliated companies

Table 6.2: 1 Important protocol violations

| Category<br>/Code | | Description |
|---|---|---|
| A | | Entrance criteria not met |
| | A1 | Inclusion criteria violated |
| | A2 | Exclusion criteria violated |
| В | | Informed consent |
| | B1 | Informed consent not available |
| | B2 | Informed consent too late |
| C | | Trial medication and randomisation |
| | C1 | Incorrect trial medication taken |
| | C2 | Randomisation not followed |
| | С3 | Non-compliance |
| | C4 | Medication code broken inappropriately |
| | C5 | Incorrect intake of trial medication |
| | C6 | Improper washout between treatments |
| D | | Concomitant medication |
| | D1 | Concomitant medication with the potential to affect the assessment of the trial medication |
| E | | Missing data |
| | E1 | Certain violations of procedures used to measure primary or secondary data |
| F | | Incorrect timing <sup>1</sup> |
| | F1 | Certain violations of time schedule used to measure primary or secondary data |
| G | | Other trial specific important violations |
| | G1 | Incorrect intake of meal |
| | G2 | PVs affecting safety and rights |

Time deviations will only be flagged as important PV, when leading to exclusion of the entire subject from an analysis set Source: 'Protocol Violation Handling Definitions' [001-MCS-50-413\_RD-01] (3)

#### PATIENT SETS ANALYSED 6.3

Treated set (TS):

This subject set includes all subjects who were documented to have received one dose of study drug.

This is the full analysis set population in the sense of ICH-E9 (1). It is used for safety analyses.

**Section 7.3 of the CTP:** Plasma concentration data and parameters of a subject will be included in the statistical pharmacokinetic analyses if they are not flagged for exclusion due to a protocol violation relevant to the evaluation of PK (to be decided no later than in the Report Planning Meeting) or due to PK non-evaluability (as revealed during data analysis, based on the criteria specified below). Exclusion of a subject's data will be documented in the CTR.

Relevant protocol violations may be:

- Incorrect trial medication taken, i.e. the subject received at least one dose of trial medication the subject was not assigned to
- Incorrect dose of trial medication taken
- *Use of restricted medications*

Plasma concentrations and/or PK parameters of a subject will be considered as nonevaluable, if for example:

- The subject experienced emesis that occurred at or before two times median  $t_{max}$  of the respective treatment (Median  $t_{max}$  is to be determined excluding the subjects experiencing emesis)
- Missing samples/concentration data at important phases of PK disposition curve
- Use of restricted comedication
- PK parameter analysis set (PKS): This subject set includes all subjects in the TS who provide at least one primary or secondary PK parameter that was not excluded according to the description above. Thus, a subject will be included in the PKS, even if he contributes only one PK parameter value for one period to the statistical assessment.

The descriptive analysis of PK concentrations will be based on the analysis data set (ADS) ADPC as described at the beginning of Section 7.

TSAP for BI Trial No: 1305-0020

Proprietary confidential information © 2018 Boehringer Ingelheim International GmbH or one or more of its affiliated companies

Table 6.3: 1 Subject sets analysed

| | Analysis se | |
|------------------------------------------------|-------------|-----|
| Class of endpoint | TS | PKS |
| Analyses of primary and secondary PK endpoints | | X |
| Safety endpoints | X | |
| Demographic/baseline endpoints | X | |
| Important protocol violations | X | |
| Disposition | X | |

### 6.5 POOLING OF CENTRES

This section is not applicable, because the study was performed in only one centre.

#### 6.6 HANDLING OF MISSING DATA AND OUTLIERS

Data of screened subjects who were withdrawn from the trial prior to first administration of any study drug will not be reported in the CTR. Handling of missing data and outliers will be performed as described in the CTP, Section 7.4.

The only exception where imputation might be necessary for safety evaluation is AE dates. Missing or incomplete AE dates are imputed according to BI standards (see 001-MCG-156 RD-01 (4)).

Missing data and outliers of PK data are handled according to BI standards (see 001-MCS-36-472 RD-01) (5).

### 6.7 BASELINE, TIME WINDOWS AND CALCULATED VISITS

The baseline value is defined as the last measurement before trial drug administration in each treatment period.

For laboratory parameters the baseline is defined as the last measurement prior to first administration of study drug.

**Section 6.1 of the CTP:** Exact times of measurements outside the permitted time windows will be documented. The acceptable time windows for screening and end of trial examination are given in the CTP Flow Chart.

TSAP for BI Trial No: 1305-0020

Proprietary confidential information © 2018 Boehringer Ingelheim International GmbH or one or more of its affiliated companies

Study measurements and assessments scheduled to occur 'before' trial medication administration on Day 1 are to be performed and completed within a 3 h-period prior to the trial drug administration and prior to predose meal intake.

The acceptable deviation from the scheduled time for post-dose vital signs, ECG and laboratory tests will be  $\pm$  30 min.

Adherence to time windows will be checked via the consistency check listings at the RPM/DBLM.

#### 7. PLANNED ANALYSIS

Safety analysis (refer to Section 7.8) will be performed by and will be presented in Sections 15.1 to 15.4 of the CTR and in Appendix 16.2 and 16.1.9.2.

Inferential statistical analyses of PK endpoints (refer to Section 7.4 and Section 7.5.2) will also be performed by and will be presented in Section 15.5 of the CTR and in Appendix 16.1.9.3.

Descriptive data analysis of PK parameters and concentrations will be performed by BI and presented in Section 15.6 of the CTR.

The format of the listings and tables will follow the standards defined in the BI corporate guideline "Reporting of Clinical Trials and Project Summaries" [001-MCG-159] (6) with the exception of those generated for PK-calculations.

The individual values of all subjects will be listed, sorted by treatment sequence, subject number, visit and actual treatment (if appropriate). The listings will be included in Appendix 16.2 of the CTR.

For end-of-text tables, the set of summary statistics for non-PK parameters is:

N number non-missing observations

arithmetic mean Mean SD standard deviation

Min minimum Median median Max maximum

For analyte concentrations as well as for all PK parameters, the following descriptive statistics will additionally be calculated:

CVarithmetic coefficient of variation

gMean geometric mean

geometric coefficient of variation gCV

P10 10th percentile 1st quartile Q1 Q3 3rd quartile P90 90th percentile

The descriptive statistics of PK parameters will be calculated using the individual values with the number of decimal places as provided by the evaluation program. Then the individual values as well as the descriptive statistics will be reported with three significant digits in the CTR.

Tabulations of frequencies for categorical data will include all possible categories and will display the number of observations in a category, as well as the percentage (%) for each

treatment group. Percentages will be rounded to one decimal place and will be based on all subjects in the respective subject set whether they have non-missing values or not. The category 'missing' will be displayed only if there are actually missing values.

Units of variables should be given in the titles or column/row descriptors in square brackets (e.g. [mg]).

### Exclusion of PK parameters

The analysis data set (ADS) ADPP contains column variables APEXC and APEXCO indicating inclusion/exclusion (APEXC) of a PK parameter and an analysis flag comment (APEXCO). All analyses based on the PKS will include parameters if they are not flagged for exclusion, that is APEXCO is equal to "Included".

## Exclusion of PK concentrations

The ADS ADPC (PK concentrations per time-point or per time-interval) contains column variables ACEXC or ACEXCO indicating inclusion/exclusion (ACEXC) of a concentration and an analysis flag comment (ACEXCO). Exclusion of a concentration depends on the analysis flag comment ACEXCO. For example, if ACEXCO is set to 'ALL CALC', the value will be excluded for all types of analyses based on concentrations. If ACEXCO is set to 'DESC STATS' the value will be excluded from descriptive evaluations per planned time point/time interval. If ACEXCO contains the addition 'TIME VIOLATION' or 'TIME DEVIATION' the value can be used for further analyses based on actual times. If ACEXCO is set to 'HALF LIFE' the value will be excluded from half-life calculation only; the value is included for all other analyses.

Further details are given in 001-MCS-36-472\_RD-01 "Noncompartmental Pharmacokinetic / Pharmacodynamic Analyses of Clinical Studies" (5) and 001-MCS-36-472\_RD-03 "Description of Analytical Transfer Files and PK/PD Data Files" (11).

#### 7.1 DEMOGRAPHIC AND OTHER BASELINE CHARACTERISTICS

Only descriptive statistics are planned for this section of the report, based on the TS.

The data will be summarised by treatment sequence and in total.

### 7.2 CONCOMITANT DISEASES AND MEDICATION

Frequency tables are planned for this section of the report, based on the TS.

Concomitant diseases will be coded using the coding system of the Medical Dictionary for Drug Regulatory Activities (MedDRA). Medications will be coded using the World Health Organization Drug Dictionary (WHO-DD). The coding version number will be displayed as a footnote in the respective output.

The diagnoses and medications will be listed. Subjects without any concomitant diagnoses or concomitant therapies should be marked with a "No" in the respective column.

The relevance of the concomitant therapies to the evaluation of PK will be decided no later than at the RPM/DBLM.

#### 7.3 TREATMENT COMPLIANCE

**Section 4.3 of the CTP:** Compliance will be assured by administration of all trial medication in the study center under supervision of the investigating physician or a designee. The measured plasma concentrations will provide additional confirmation of compliance.

It is not intended to list the compliance separately. Any deviations from complete intake will be addressed in the RPM/DBLM (cf. TSAP <u>Section 6.2</u>) and described in the CTR.

### 7.4 PRIMARY ENDPOINTS

Relative bioavailability is to be determined on the basis of the primary and secondary pharmacokinetic endpoints (see Section 5.1).

The PK endpoints will be log-transformed (natural logarithm) prior to fitting the ANOVA model (see below).

#### Primary analysis

The statistical model used for the analysis of primary and secondary PK endpoints will be an ANOVA (analysis of variance) model on the logarithmic scale (see below).

**Section 7.3.1 of the CTP:** This model will include effects accounting for the following sources of variation: 'sequence', 'subjects within sequences', 'period' and 'treatment'. The effect 'subjects within sequences' will be considered as random, whereas the other effects will be considered as fixed. The model is described by the following equation:

$$y_{ijkm} = \mu + \zeta_i + s_{im} + \pi_i + \tau_k + e_{ijkm}$$
, where

 $y_{ijkm} = logarithm \ of \ response \ (AUC_{0-tz}, C_{max}, AUC_{0-\infty})$  measured on subject m in sequence i receiving treatment k in period j,

 $\mu$  = the overall mean,

$$\zeta_i = the i^{th}$$
 sequence effect,  $i = 1, 2$ 

 $s_{im}$  = the effect associated with the  $m^{th}$  subject in the  $i^{th}$  sequence, m = 1, 2, ..., 6, i=1, 2

$$\pi_i = the j^{th} period effect, j = 1, 2$$

$$\tau_k$$
 = the  $k^{th}$  treatment effect,  $k = 1, 2$ 

 $e_{ijkm}$  = the random error associated with the  $m^{th}$  subject in sequence i who received treatment k in period j.

The difference between the expected means for test treatments (tablets under fed conditions, T) and reference treatment (tablets under fasted conditions, R) ln(T)-ln(R), will be estimated by the difference in the corresponding Least Square Means (point estimate) and two-sided 90% confidence intervals based on the t-distribution will be computed. These quantities will then be back-transformed to the original scale to give the point estimator (geometric mean) and interval estimates for the ratio between response under test and response under reference.

The analysis will be accomplished by using the XPKISTAT macro, based on PKS (design BWC).

#### 7.5 SECONDARY ENDPOINTS

### 7.5.1 Key secondary endpoints

This section is not applicable as no key secondary endpoint has been specified in the protocol.

### 7.5.2 Secondary endpoints

The secondary PK endpoint  $AUC_{0-\infty}$  will be assessed using the same methods as described for the primary endpoints but will not be interpreted in a confirmatory sense.

### 7.7 EXTENT OF EXPOSURE

Descriptive statistics are planned for this section of the report based on the TS. The date and time of drug administration will be listed for each subject.

#### 7.8 SAFETY ANALYSIS

All safety analyses will be performed on the TS.

If not stated otherwise, the safety results will be sorted by actual treatment.

The safety data for treated subjects who failed to complete the study (dropouts or withdrawals) will be reported as far as their data are available. All withdrawals will be documented and the reason for withdrawal recorded.

#### 7.8.1 Adverse events

AEs will be coded with the most recent version of MedDRA.

The analyses of AEs will be descriptive in nature and will be based on BI standards as presented in the corporate guideline: "Analysis and Presentation of Adverse Event Data from Clinical Trials" [001-MCG-156] (8).

The standard AE analyses will be based on the number of subjects with AEs (and not on the number of AEs).

For analysis, multiple AE occurrence data on the CRF will be collapsed into an AE provided that all of the following applies:

- All AE attributes are identical (LLT, intensity, action taken, therapy required, seriousness, reason for seriousness, relationship, outcome, AE of special interest)
- The occurrences were time-overlapping or time-adjacent (time-adjacency of 2 occurrences is given if the second occurrence started within one hour after end of the first occurrence).

For further details on summarization of AE data, please refer to [001-MCG-156] (8,4).

**Section 5.2.2.1 of the CTP:** *The following are considered as AESIs in this trial:* 

- Hepatic injury, as defined by the following alterations of hepatic laboratory parameters:
  - o an elevation of AST and/or ALT  $\geq$ 3-fold ULN combined with an elevation of total bilirubin  $\geq$ 2-fold ULN measured in the same blood sample, and/or
  - o marked peak aminotransferase (ALT, and/or AST) elevations  $\geq$ 10 fold ULN

These lab findings constitute a hepatic injury alert and the patients showing these lab abnormalities need to be followed up according to the 'DILI checklist' provided in the ISF. In case of clinical symptoms of hepatic injury (icterus, unexplained encephalopathy, unexplained coagulopathy, right upper quadrant abdominal pain, etc.) without lab results (ALT, AST, total bilirubin) available, the Investigator should make sure these parameters are analyzed, if necessary in an unscheduled blood test. Should the results meet the criteria of hepatic injury alert, the procedures described in the DILI checklist should be followed.

With the exception of DILI, no AESIs have been defined for this trial.

The analysis of adverse events will be based on the concept of treatment emergent adverse events.

**Section 5.2.2.2 of the CTP:** The Residual Effect Period (REP) for BI 1015550, when measurable drug levels or PD effects are still likely to be present, is defined as after the last administration of BI 1015550. Therefore, all AEs which occurred through the treatment phase and throughout the REP will be considered as on treatment [...].

All adverse events occurring before first drug administration will be assigned to 'screening', those between intake of trial medication and end of the will be assigned to the corresponding treatment ('on treatment'). AEs occurring after the REP but prior to next drug administration or termination date will be assigned to 'follow-up'. The follow-up will be summarized according to previous treatment.

According to ICH E3 (9), AEs classified as 'other significant' need to be reported and will include those non-serious and non-significant adverse events with

- (i) 'action taken = discontinuation' or 'action taken = reduced', or
- (ii) marked haematological and other lab abnormalities or lead to significant concomitant therapy as identified by the Clinical Monitor/Investigator at the Report Planning Meeting.

An overall summary of AEs (including AESIs) will be presented.

The frequency of subjects with AEs will be summarised by treatment, primary system organ class (SOC) and preferred term (PT). Separate tables will be provided for subjects with other significant AEs according to ICH E3 (9), for subjects with serious AEs, for subjects with drug-related AEs, for subjects with drug related serious adverse events and for subjects with AESIs.

The SOC and PTs will be sorted by frequency. The MedDRA version number will be displayed as a footnote in the respective output.

In addition, for disclosure of AE data on ClinicalTrials.gov, frequencies of subjects with nonserious AEs that had an incidence of > 5% (in preferred term) for at least one treatment will be summarised by treatment, primary SOC and PT.

For disclosure of adverse events on EudraCT, additional information not included in a standard AE analysis will be performed. The following three entries will be created:

- Adverse Events per arm for disclosure on EudraCT
- Non-serious Adverse Events for disclosure on EudraCT
- Serious Adverse Events for disclosure on EudraCT

#### 7.8.2 Laboratory data

The analyses of laboratory data will be descriptive in nature and will be based on BI standards [001-MCG-157] (10).

Laboratory data will be analysed qualitatively via comparison of laboratory data to their reference ranges. Values outside the reference range as well as values defined as clinically relevant will be highlighted in the data listings.

Possibly clinically significant abnormal laboratory values are only those identified either in the Investigator's comments on the CRF or at the RPM/DBLM at the latest. It is the investigator's responsibility to decide whether a lab value is clinically significant abnormal or not. Standard or project-specific rules for flagging clinically significant values will not be applied in this study.

#### 7.8.3 Vital signs

Descriptive statistics over time including change from baseline will be performed for vital signs (blood pressure and pulse rate).

#### 7.8.4 **ECG**

ECG recordings will be checked by the investigator for pathological results. Clinically relevant abnormal findings for ECG will be listed under 'Relevant Medical History / Baseline Conditions' (when they occurred during screening) or will be reported as AEs (when they occurred during treatment).

#### 7.8.5 **Others**

This section is not applicable as no other variables have been specified in the protocol.

### 8. REFERENCES

- 1 *CPMP/ICH/363/96:* "Statistical Principles for Clinical Trials", ICH Guideline Topic E9, Note For Guidance on Statistical Principles for Clinical Trials, current version.
- 2 001-MCS-50-413\_RD-02: "Important Manual Protocol Violations Spreadsheet", current version, IDEA for CON.
- 3 001-MCS-50-413\_RD-01: "Protocol Violation Handling Definitions", current version, IDEA for CON.
- 4 001-MCG-156\_RD-01: "Handling of Missing and Incomplete AE Dates", current version; IDEA for CON.
- 5 001-MCS-36-472\_RD-01: "Noncompartmental Pharmacokinetic/Pharmacodynamic Analyses of Clinical Studies", current version; IDEA for CON.
- 6 001-MCG-159: "Reporting of Clinical Trials and Project Summaries", current version; IDEA for CON.
- 7 001-MCS-36-472: "Standards and processes for analyses performed within Clinical Pharmacokinetics/Pharmacodynamics", current version; IDEA for CON.
- 8 001-MCG-156: "Analysis and Presentation of Adverse Event Data from Clinical Trials", current version; IDEA for CON.
- 9 *CPMP/ICH/137/95*: "Structure and Content of Clinical Study Reports", ICH Guideline Topic E3; Note For Guidance on Structure and Content of Clinical Study Reports, current version.
- 10 001-MCG-157: "Handling, Display and Analysis of Laboratory Data", current version; IDEA for CON.
- 11 001-MCS-36-472\_RD-03: "Description of Analytical Transfer Files and PK/PD Data Files", current version; IDEA for CON.

TSAP for BI Trial No: 1305-0020 

Proprietary confidential information © 2018 Boehringer Ingelheim International GmbH or one or more of its affiliated companies

TSAP for BI Trial No: 1305-0020 

Proprietary confidential information © 2018 Boehringer Ingelheim International GmbH or one or more of its affiliated companies

#### **10. HISTORY TABLE**

Table 10: 1 History table

| Version | Date | Author | Sections | Brief description of change |
|---|---|---|---|---|
| | (DD-MMM-YY) | | changed | |
| Final | 19-JAN-18 | | None | This is the final TSAP without any modification |